CLINICAL TRIAL: NCT03443726
Title: Is the Direct Inferior Alveolar Nerve Block Required for Third Lower Molar Extraction?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Rui Figueiredo, Professor, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UBarcelonaOralSurgery1
Record Dates: First submitted 2017-12-20; First posted 2018-02-23 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Tooth Extraction; Dental Anesthesia
Keywords: Lower third molar extraction; Infiltration anesthesia; Articaine
MeSH Terms: interventions — Carticaine; Epinephrine

STUDY DESIGN:
Intervention Model Description: * Control group: inferior alveolar nerve block with 1.8 cc of 4% articaine 1:100.000 epinephrine and 1.8 cc of the same anesthetic for the buccal nerve block.
  * Test group: infiltration anesthesia buccaly between first and second mandibular molar with 3.6 cc of 4% articaine 1:100.000 epinephrine and 0.6 cc ligually to the third molar using the same anesthetic.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: * The participant is not told which technique will be used on him/her.
  * Surgeon does not know the anesthetic technique used to numb the third molar.
  * When the statistician and primary investigator receive the collected data to be analyzed, the techniques are labeled 1 and 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Infiltrative technique (Experimental): Patients in this arm will have buccal and lingual infiltrative anesthesia with 4% articaine 1:100.000 epinephrine for third molar extraction.
  Interventions: Procedure: Infiltrative technique; Drug: 4% articaine 1:100.000 epinephrine; Procedure: Third molar extraction
- Nerve block technique (Active Comparator): Patients in this arm will have inferior alveolar nerve and buccal nerve block with 4% articaine 1:100.000 epinephrine for third molar extraction.
  Interventions: Procedure: Nerve block technique; Drug: 4% articaine 1:100.000 epinephrine; Procedure: Third molar extraction

INTERVENTIONS:
Procedure: Nerve block technique — Inferior alveolar nerve block with 1.8 cc of 4% articaine 1:100.000 epinephrine and 1.8 cc of the same anesthetic for the buccal nerve for third molar extraction.
  Other Names: Standard intervention
  Arms: Nerve block technique
Procedure: Infiltrative technique — Infiltrative anesthesia buccally between first and second mandibular molar with 3.6 cc of 4% articaine 1:100.000 epinephrine and 0.6 cc lingually to the third molar using the same anesthetic solution.
  Other Names: Experimental intervention
  Arms: Infiltrative technique
Drug: 4% articaine 1:100.000 epinephrine — Articaine in a 4% solution with epinephrine 1:100,000 (Artinibsa; Inibsa Dental, Lliçà de Vall, Spain)
Procedure: Third molar extraction — Third molar extraction under local anesthesia.

SUMMARY:
This study is a Randomized Controlled Trial (RCT) which objective is to compare the effectiveness, efficacy and complication associated to an infiltrative anesthetic technique for the removal of lower third molars comparing it to the standard inferior alveolar nerve block using 4% articaine 1:100.000 epinephrine.

DETAILED DESCRIPTION:
The objective is to compare the anesthetic efficacy of an infiltrative anesthetic technique placed buccally between the first and second mandibular molars plus infiltration of the third molar's lingual mucosa with the direct inferior alveolar nerve block plus buccal nerve block for the extraction of lower wisdom teeth. All using 4% articaine 1:100.000 epinephrine. The first technique is to be referred as Alternative Technique (A.T.) and the second Standard Technique (S.T.) The study is being conducted at the Hospital Odontològic Universitat de Barcelona (Campus de Bellvitge) and is being carried out by members of the Oral Surgery and Implantology Master's program of the University of Barcelona.

The sample (110 patients) consists of patients in need of lower third molar extraction. All of them are being properly informed about the study according to the Comité Ético (CEIC) del Hospital Odontològic Universitat de Barcelona guidelines, and informed consent must be signed prior to the interventions. All patients derive from the Institut Català de la Salut-Consorci Sanitari.

The materials used are 1.8cc carpules of 4% articaine and 1:100.000 epinephrine, dental anesthetic syringe, dental anesthetic needles of 35 mm 27G and 25 mm 27G as well as all the documents necessary for data collection.

The determinations to be done are the pulpal anesthetic efficacy (in seconds, using a pulpometer), chin and tongue numbness (patient reported, measured in seconds), need for supplemental anesthesia, comfort (pain experienced during the punctions and during and after surgery), morbility (cramp sensation in the tongue or lip when performing the anesthetic technique, local and/or systemic complications).

ELIGIBILITY:
Inclusion Criteria:

* Lower third molars in any position (in accordance to Pell and Gregory and Winter classification) in need of extraction.
* Healthy patients and patients with mild systemic disease without substantive functional limitations (ASA I-II).
* Absence of acute infection in the third molar area.
* Adequate intellectual capacity for understanding the nature and purpose of the study and fill the informed consent and questionaries appropriately.

Exclusion Criteria:

* History of recent trauma in the maxillofacial area.
* Articaine or lidocaine allergy.
* Presence of a systemic pathology that contraindicates the use of local anesthetics with vasopressors.
* Acute infection in the third molar area (in the las 30 days).
* Surgeries taking more than 60 minutes (automatic dropout).
* Unwillingness to participate or continue participating in the study.
* A score equal or superior to 13 points in the Corah´s anxiety test.
* Third molars in ectopic position.
* Caries on the third molar.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-06-10 (Actual); Primary Completion 2018-11-10 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Need for supplemental anesthesia [Efficacy] | At the end of surgery (≤60 minutes after pulpal anesthesia is achieved)
  Using a questionnaire filled by the surgeon at the end of surgery. Need for supplemental anesthesia (yes/no)

SECONDARY OUTCOMES:
Local anesthetic injection pain | After local anesthetic injection (minute 0)
  Measured by a 100 mm Visual Analog Scale (VAS) Range: 0 mm [No pain. Best outcome] to 100 mm [Worst pain. Worst outcome]
Morbidity | After local anesthetic injection (minute 0)
  Using a questionnaire. Electrical shock sensation affecting lower lip and/or tongue (yes/no).
Latency | After anesthetic injection (approximately 0 to 360 seconds)
  Time elapsed from anesthetic injection to numbness of tongue and lower lip (Vicent's sign) reported by the patient (seconds).
Pulpal anesthesia | Minute 1 (after Vincent's sign is achieved)
  Using an electronic pulp tester placed on the mesiobuccal cusp tip of ipsilateral lower second molar.
  No response at 80 units.
Pulpal anesthesia | Minute 1.5 (after Vincent's sign is achieved)
  Using an electronic pulp tester placed on the mesiobuccal cusp tip of ipsilateral lower second molar.
  No response at 80 units.
Pulpal anesthesia | Minute 2 (after Vincent's sign is achieved)
  Using an electronic pulp tester placed on the mesiobuccal cusp tip of ipsilateral lower second molar.
  No response at 80 units.
Pulpal anesthesia | Minute 2.5 (after Vincent's sign is achieved)
  Using an electronic pulp tester placed on the mesiobuccal cusp tip of ipsilateral lower second molar.
  No response at 80 units.
Pulpal anesthesia | Minute 3 (after Vincent's sign is achieved)
  Using an electronic pulp tester placed on the mesiobuccal cusp tip of ipsilateral lower second molar.
  No response at 80 units.
Pulpal anesthesia | Minute 3.5 (after Vincent's sign is achieved)
  Using an electronic pulp tester placed on the mesiobuccal cusp tip of ipsilateral lower second molar.
  No response at 80 units.
Pulpal anesthesia | Minute 4 (after Vincent's sign is achieved)
  Using an electronic pulp tester placed on the mesiobuccal cusp tip of ipsilateral lower second molar.
  No response at 80 units.
Pulpal anesthesia | Minute 4.5 (after Vincent's sign is achieved)
  Using an electronic pulp tester placed on the mesiobuccal cusp tip of ipsilateral lower second molar.
  No response at 80 units.
Pulpal anesthesia | Minute 5 (after Vincent's sign is achieved)
  Using an electronic pulp tester placed on the mesiobuccal cusp tip of ipsilateral lower second molar.
  No response at 80 units.
Pulpal anesthesia | Minute 5.5 (after Vincent's sign is achieved)
  Using an electronic pulp tester placed on the mesiobuccal cusp tip of ipsilateral lower second molar.
  No response at 80 units.
Pulpal anesthesia | Minute 6 (after Vincent's sign is achieved)
  Using an electronic pulp tester placed on the mesiobuccal cusp tip of ipsilateral lower second molar.
  No response at 80 units.
Surgery pain | At the end of surgery (≤60 minutes after pulpal anesthesia is achieved)
  Measured by a 100 mm Visual Analog Scale (VAS) Range: 0 mm [No pain. Best outcome] to 100 mm [Worst pain. Worst outcome]
Post operative pain | 2 hours
  Measured by a 100 mm Visual Analog Scale (VAS) Range: 0 mm [No pain. Best outcome] to 100 mm [Worst pain. Worst outcome]
Post operative pain | 6 hours
  Measured by a 100 mm Visual Analog Scale (VAS) Range: 0 mm [No pain. Best outcome] to 100 mm [Worst pain. Worst outcome]
Post operative pain | 12 hours
  Measured by a 100 mm Visual Analog Scale (VAS) Range: 0 mm [No pain. Best outcome] to 100 mm [Worst pain. Worst outcome]
Post operative pain | 24 hours
  Measured by a 100 mm Visual Analog Scale (VAS) Range: 0 mm [No pain. Best outcome] to 100 mm [Worst pain. Worst outcome]
Post operative pain | Day 1
  Measured by a 100 mm Visual Analog Scale (VAS) Range: 0 mm [No pain. Best outcome] to 100 mm [Worst pain. Worst outcome]
Post operative pain | Day 2
  Measured by a 100 mm Visual Analog Scale (VAS) Range: 0 mm [No pain. Best outcome] to 100 mm [Worst pain. Worst outcome]
Post operative pain | Day 3
  Measured by a 100 mm Visual Analog Scale (VAS) Range: 0 mm [No pain. Best outcome] to 100 mm [Worst pain. Worst outcome]
Post operative pain | Day 4
  Measured by a 100 mm Visual Analog Scale (VAS) Range: 0 mm [No pain. Best outcome] to 100 mm [Worst pain. Worst outcome]
Post operative pain | Day 5
  Measured by a 100 mm Visual Analog Scale (VAS) Range: 0 mm [No pain. Best outcome] to 100 mm [Worst pain. Worst outcome]
Post operative pain | Day 6
  Measured by a 100 mm Visual Analog Scale (VAS) Range: 0 mm [No pain. Best outcome] to 100 mm [Worst pain. Worst outcome]
Post operative pain | Day 7
  Measured by a 100 mm Visual Analog Scale (VAS) Range: 0 mm [No pain. Best outcome] to 100 mm [Worst pain. Worst outcome]
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Day 7
  Using a questionnaire filled by the surgeon at the end of study visit. Pruritus, nausea, vomiting, bleeding, anesthesia of the mouth, difficulty breathing, drowsiness, headache, sweating, palpitations, skin rash, difficult deglutition and dysarthria during the follow-up period (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Rui Figueiredo, DDS, MS, PhD, Study Director — University of Barcelona; Eduard Valmaseda-Castellon, DDS, MS. PhD, Study Chair — University of Barcelona; Stavros J Sofos, DDS, MS., Principal Investigator — University of Barcelona, Nova Southeastern University.; Leonardo Berini-Aytes, MD, DDS, PhD, Principal Investigator — University of Barcelona; Octavi Camps-Font, DDS, MS, Principal Investigator — University of Barcelona
Locations (1):
- University of Barcelona, L'Hospitalet de Llobregat, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Berini Aytés L, Gay Escoda C, Uribarri A. Técnica de anestesia por bloqueo en la mandíbula. En: Berini Aytés L, Gay Escoda C. (eds.). Anestesia Odontológica, 3o ed. Madrid: Avances médico- dentales; 2005. p. 253-79.
- [Background] Meechan JG. The use of the mandibular infiltration anesthetic technique in adults. J Am Dent Assoc. 2011 Sep;142 Suppl 3:19S-24S. doi: 10.14219/jada.archive.2011.0343. PMID 21881058
- [Background] Kanaa MD, Whitworth JM, Corbett IP, Meechan JG. Articaine and lidocaine mandibular buccal infiltration anesthesia: a prospective randomized double-blind cross-over study. J Endod. 2006 Apr;32(4):296-8. doi: 10.1016/j.joen.2005.09.016. Epub 2006 Feb 17. PMID 16554198
- [Background] Kanaa MD, Whitworth JM, Corbett IP, Meechan JG. Articaine buccal infiltration enhances the effectiveness of lidocaine inferior alveolar nerve block. Int Endod J. 2009 Mar;42(3):238-46. doi: 10.1111/j.1365-2591.2008.01507.x. PMID 19228214
- [Background] Corbett IP, Kanaa MD, Whitworth JM, Meechan JG. Articaine infiltration for anesthesia of mandibular first molars. J Endod. 2008 May;34(5):514-8. doi: 10.1016/j.joen.2008.02.042. PMID 18436027
- [Background] Meechan JG. Infiltration anesthesia in the mandible. Dent Clin North Am. 2010 Oct;54(4):621-9. doi: 10.1016/j.cden.2010.06.003. PMID 20831926
- [Background] Pogrel MA, Thamby S. Permanent nerve involvement resulting from inferior alveolar nerve blocks. J Am Dent Assoc. 2000 Jul;131(7):901-7. doi: 10.14219/jada.archive.2000.0308. PMID 10916328
- [Background] Renton T, Adey-Viscuso D, Meechan JG, Yilmaz Z. Trigeminal nerve injuries in relation to the local anaesthesia in mandibular injections. Br Dent J. 2010 Nov;209(9):E15. doi: 10.1038/sj.bdj.2010.978. PMID 21072069
- [Background] Hillerup S, Jensen R. Nerve injury caused by mandibular block analgesia. Int J Oral Maxillofac Surg. 2006 May;35(5):437-43. doi: 10.1016/j.ijom.2005.10.004. Epub 2005 Dec 15. PMID 16343853
- [Background] Delgado-Molina E, Tamarit-Borras M, Berini-Aytes L, Gay-Escoda C. Comparative study of two needle models in terms of deflection during inferior alveolar nerve block. Med Oral Patol Oral Cir Bucal. 2009 Sep 1;14(9):e440-4. PMID 19718006
- [Background] Hillerup S, Jensen RH, Ersboll BK. Trigeminal nerve injury associated with injection of local anesthetics: needle lesion or neurotoxicity? J Am Dent Assoc. 2011 May;142(5):531-9. doi: 10.14219/jada.archive.2011.0223. PMID 21531935
- [Background] Moore PA, Haas DA. Paresthesias in dentistry. Dent Clin North Am. 2010 Oct;54(4):715-30. doi: 10.1016/j.cden.2010.06.016. PMID 20831934
- [Background] Garisto GA, Gaffen AS, Lawrence HP, Tenenbaum HC, Haas DA. Occurrence of paresthesia after dental local anesthetic administration in the United States. J Am Dent Assoc. 2010 Jul;141(7):836-44. doi: 10.14219/jada.archive.2010.0281. PMID 20592403
- [Background] Gaffen AS, Haas DA. Retrospective review of voluntary reports of nonsurgical paresthesia in dentistry. J Can Dent Assoc. 2009 Oct;75(8):579. PMID 19840499
- [Background] Malamed SF, Gagnon S, Leblanc D. Articaine hydrochloride: a study of the safety of a new amide local anesthetic. J Am Dent Assoc. 2001 Feb;132(2):177-85. doi: 10.14219/jada.archive.2001.0152. PMID 11217590
- [Background] Gay Escoda C, Berini Aytés. Técnicas anestésicas en Cirugía Bucal. En: Tratado de Cirugía Bucal. Madrid: Ergon; 2004. p. 155-98
- [Background] Torrente-Castells E, Gargallo-Albiol J, Rodriguez-Baeza A, Berini-Aytes L, Gay-Escoda C. Necrosis of the skin of the chin: a possible complication of inferior alveolar nerve block injection. J Am Dent Assoc. 2008 Dec;139(12):1625-30. doi: 10.14219/jada.archive.2008.0104. PMID 19047668
- [Background] Brandt RG, Anderson PF, McDonald NJ, Sohn W, Peters MC. The pulpal anesthetic efficacy of articaine versus lidocaine in dentistry: a meta-analysis. J Am Dent Assoc. 2011 May;142(5):493-504. doi: 10.14219/jada.archive.2011.0219. PMID 21531931
- [Background] Meechan JG, Jaber AA, Corbett IP, Whitworth JM. Buccal versus lingual articaine infiltration for mandibular tooth anaesthesia: a randomized controlled trial. Int Endod J. 2011 Jul;44(7):676-81. doi: 10.1111/j.1365-2591.2011.01878.x. Epub 2011 Mar 30. PMID 21447137
- [Background] El-Kholey KE. Infiltration anesthesia for extraction of the mandibular molars. J Oral Maxillofac Surg. 2013 Oct;71(10):1658.e1-5. doi: 10.1016/j.joms.2013.06.203. PMID 24040947
- [Background] Montserrat-Bosch M, Figueiredo R, Nogueira-Magalhaes P, Arnabat-Dominguez J, Valmaseda-Castellon E, Gay-Escoda C. Efficacy and complications associated with a modified inferior alveolar nerve block technique. A randomized, triple-blind clinical trial. Med Oral Patol Oral Cir Bucal. 2014 Jul 1;19(4):e391-7. doi: 10.4317/medoral.19554. PMID 24608204